CLINICAL TRIAL: NCT00122447
Title: CVD Risk and Prevention in Early Glucose Intolerance
Brief Title: Cardiovascular Disease (CVD) Risk and Prevention in Early Glucose Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Daiichi Sankyo (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Dr. Mary Rhee, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00000749; UL1RR025008 (NIH); Sankyo CS-866 (Other: Daiichi Sankyo); 1K23DK070715-01A1 (NIH)
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Impaired Glucose Tolerance; Prediabetic State
Keywords: Prediabetic state; Cardiovascular disease; Diabetes; Glucose intolerance
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State; Cardiovascular Diseases; Diabetes Mellitus | interventions — Aspirin; Thioctic Acid; olmesartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Anti-inflammatory agent (Active Comparator): Aspirin (ASA)
  Interventions: Drug: Aspirin
- Angiotensin receptor blocker (ARB) (Active Comparator): Olmesartan (ARB)
  Interventions: Drug: Olmesartan
- Antioxidant (Active Comparator): Alpha lipoic acid (ALA)
  Interventions: Drug: Alpha lipoic acid
- Placebo (Placebo Comparator): Aspirin placebo once a day Olmesartan placebo once a day Alpha lipoic acid placebo twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 325 mg PO QD
  Other Names: Bayer aspirin
  Arms: Anti-inflammatory agent
Drug: Alpha lipoic acid — 600 mg PO BID
  Arms: Antioxidant
Drug: Olmesartan — 40 mg PO QD
  Other Names: Benicar
  Arms: Angiotensin receptor blocker (ARB)
Drug: Placebo — Identical placebo for each active comparator:
  placebo aspirin 325 mg PO QD; placebo for alpha lipoic acid 600 mg PO BID; placebo for olmesartan 40 mg PO QD
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether cardiovascular disease (CVD) risk markers, β-cell function, and insulin sensitivity can be improved by targeting mechanisms of both diabetes and CVD - using an antioxidant, an angiotensin II receptor blocker (ARB), or an anti-inflammatory agent - in patients with impaired glucose tolerance (IGT) in a randomized, controlled trial.

DETAILED DESCRIPTION:
Diabetes is a common, major health problem in the United States, and it significantly increases the risk of developing heart disease, which is the leading cause of death. Research studies have shown that the risk of heart disease is increased, even in the "pre-diabetes" or impaired glucose tolerance (IGT) stage, before the onset of true diabetes. While many studies have shown that aggressive management of diabetes lowers the risk of heart disease, at the present time, it is not known how best to treat patients with impaired glucose tolerance (pre-diabetes) to prevent the development of heart disease. It is also not known where in the range of blood sugar levels risk begins to increase. The purpose of this study is to determine:

* whether medications, which target pathways involved in the development of heart disease, can decrease the risk of heart disease in individuals with impaired glucose tolerance; and
* whether a "high" blood sugar level measured one hour after drinking a standard high-sugar drink is associated with an increased risk of heart disease even in individuals who have no evidence of diabetes or pre-diabetes.

The purpose of Aim 1 of this study is to determine whether medications, which target pathways involved in the development of heart disease, can decrease the risk of heart disease in individuals with impaired glucose tolerance. One hundred-twenty volunteers with impaired glucose tolerance and 30 volunteers with normal glucose tolerance (normal blood sugars after ingesting a standard high-sugar drink) will be recruited from the "Screening for Impaired Glucose Tolerance" (SIGT) study. The 30 volunteers with normal glucose tolerance will not take any study medication, but will undergo medical testing to determine their risk of heart disease at the beginning of the study, after which their participation in the study will be complete. The 120 volunteers with impaired glucose tolerance will be randomly assigned to one of four medications to be taken over a one-year period:

* alpha lipoic acid (an antioxidant, dietary supplement);
* olmesartan (a drug used to treat high blood pressure);
* aspirin (an anti-inflammatory drug); and
* placebo (an inactive, "dummy" pill).

Subjects with impaired glucose tolerance will undergo medical testing to determine their risk of heart disease at the beginning of the study (before beginning study medications), after 3 months of intervention, and again at the end of the study (12 months after enrollment). Test results will be compared between the subjects taking each of the active medications and those taking placebo, to determine if the medications lead to a significant reduction in the risk for the development of heart disease. The medical tests used in this study are currently used in medical practice, and include blood and urine specimens, ultrasound testing of the artery at the arm, and an insulin sensitivity test (test of how effectively the body uses sugar). All visits and tests will be conducted in the General Clinical Research Centers of Emory University Hospital and Grady Memorial Hospital.

The purpose of Aim 2 of this study is to determine whether a "high" blood sugar level measured one hour after drinking a standard high-sugar drink (1-hour blood sugar level) is associated with an increased risk of heart disease even in individuals who have no evidence of diabetes or pre-diabetes. Seventy-five volunteers with normal glucose tolerance (normal blood sugars after ingesting a standard high-sugar drink) will be recruited from the SIGT study, as well as 15 subjects with impaired glucose tolerance and 15 with diabetes. The subjects with normal glucose tolerance will be grouped into those with "low", "middle", and "high" 1-hour blood sugar levels. All subjects will undergo medical testing (as in Aim 1 above) to determine their risk of heart disease. Test results of subjects with "low", "middle", and "high" 1-hour blood sugar levels will be compared against one another, as well as against those of subjects with IGT and diabetes. If subjects with normal glucose tolerance but "high" 1-hour blood sugar levels are found to have increased risk for heart disease compared to those with "low" 1-hour blood sugar levels, then the 1-hour blood sugar levels may provide important information regarding an increased risk of heart disease even in individuals with normal glucose tolerance but "high" 1-hour blood sugar levels - a population which otherwise would not be identified with the current standard tests used for the diagnosis of diabetes and pre-diabetes.

Over 40 million Americans have pre-diabetes (impaired glucose tolerance), which is associated with an increased risk of the development of both diabetes and heart disease. Findings from these studies will provide important insights into the pathways that lead to the development of heart disease related to pre-diabetes, prevention of heart disease in the pre-diabetic population, and identification of individuals at high risk for heart disease earlier in their natural history - even before the onset of pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance

Exclusion Criteria:

* Diagnosis of diabetes
* Taking an ACE inhibitor (ACE-I), angiotensin II receptor blocker (ARB), or aspirin
* Have systolic blood pressure >140 mm Hg
* Have a chronic inflammatory disorder (i.e. rheumatoid arthritis, inflammatory bowel disease, sinusitis)
* Vascular disease (cardiac, peripheral, cerebral)
* Renal insufficiency or hepatic abnormalities
* Gastrointestinal bleeding (defined as gastric or duodenal ulcer, hematemesis, and/or blood in the stool) or significant other upper gastrointestinal problems (i.e. gastritis) within the previous 6 months
* Anemia or a history of bleeding disorder
* Have a history of ARB or aspirin allergy
* Have the syndrome of asthma, rhinitis, and nasal polyps
* Have other medical problems which would preclude taking potential study medications for 12 months
* Are pregnant or have a positive pregnancy test
* Are breast feeding
* Are unable or unwilling to tolerate having one catheter in each arm for 4 hours
* Have health status such that the envisioned blood sampling would confer a physiologic risk
* Have other physical, social, or behavioral problems which would decrease the likelihood that they would remain in the study for 12 months
* Do not appear capable of giving informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Rhee, MD, MS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 266 subjects with IGT were contacted: 121 refused, 63 ineligible, 84 screened/enrolled.
  Among the 84 enrolled subjects:
  1 was withdrawn, 13 dropped out before randomization, 70 were randomized (17 alpha lipoic acid, 18 aspirin, 18 olmesartan, 17 placebo).
  After randomization, 10 dropped out, and 3 were withdrawn.
Groups:
- Aspirin (ASA) 325 mg PO Once Daily: Anti-inflammatory agent
- Olmesartan (ARB) 40 mg PO Once Daily: Angiotensin receptor blocker (ARB)
- Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily: Antioxidant
- Placebo: Aspirin placebo PO once a day Olmesartan placebo PO once a day Alpha lipoic acid placebo PO twice a day
Period: Overall Study
Arm/Group | Aspirin (ASA) 325 mg PO Once Daily | Olmesartan (ARB) 40 mg PO Once Daily | Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily | Placebo
Started | 18 | 18 | 17 | 17
Completed | 17 | 13 | 16 | 14
Not Completed | 1 | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin (ASA) 325 mg PO Once Daily | Olmesartan (ARB) 40 mg PO Once Daily | Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.8) | 55.2 (8.5) | 52.4 (7.0) | 51.3 (11.7) | 52.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 10 | 6 | 39
  Male | 5 | 8 | 7 | 11 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 13 | 12 | 10 | 14 | 49
  White | 5 | 6 | 7 | 3 | 21

OUTCOME MEASURES:

1. Secondary Outcome: AIM 1: Change in hsCRP (High Sensitivity C-reactive Peptide) Level
Description: Inflammatory marker
Time Frame: 12 months of intervention
Population: Based on the number of subjects who completed 12 months of intervention and testing
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Aspirin (ASA) 325 mg PO Once Daily | Olmesartan (ARB) 40 mg PO Once Daily | Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 10
mg/L | -1.27 (0.86) | -2.34 (1.1) | 0.23 (0.70) | 0.32 (0.56)
Statistical Analysis 1: Comparison: Aspirin (ASA) 325 mg PO Once Daily vs Placebo; Test type: Superiority or Other; p = 0.449, Regression, Linear — Association between treatment arm, compared to placebo, on change in hsCRP from baseline to 12 months of intervention, adjusted for age, sex, and race; Slope = -0.941, 95% CI 2-sided [-3.435 to 1.552], Standard Error of Mean 1.229
Statistical Analysis 2: Comparison: Olmesartan (ARB) 40 mg PO Once Daily vs Placebo; Test type: Superiority or Other; p = 0.034, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -2.677, 95% CI 2-sided [-5.133 to -0.221], Standard Error of Mean 1.211
Statistical Analysis 3: Comparison: Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily vs Placebo; Test type: Superiority or Other; p = 0.943, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = 0.088, 95% CI 2-sided [-2.367 to 2.542], Standard Error of Mean 1.210

2. Primary Outcome: AIM 1: Change in Flow Mediated Dilation (FMD) (%)
Description: Surrogate measure of endothelial function defined as the percent change in dilation of the brachial artery after cuff compression of arm compared to before cuff compression
Time Frame: 12 months of intervention
Population: Based on the number of subjects who completed 12 months of intervention and testing
Measure: Mean (Standard Deviation); unit: percentage of arterial dilation change
Arm/Group | Aspirin (ASA) 325 mg PO Once Daily | Olmesartan (ARB) 40 mg PO Once Daily | Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily | Placebo
Number analyzed (Participants) | 17 | 13 | 15 | 13
percentage of arterial dilation change | -0.0012 (0.030) | 0.018 (0.032) | 0.014 (0.034) | 0.0053 (0.030)
Statistical Analysis 1: Comparison: Aspirin (ASA) 325 mg PO Once Daily vs Placebo; Null hypothesis: no difference between active treatment group compared to placebo; Test type: Superiority or Other; p = 0.943, Regression, Linear — Association between treatment arm, compared to placebo, on change in FMD from baseline to 12 months of intervention, adjusted for age, sex, race, and LDL-cholesterol; Slope = -0.001, 95% CI 2-sided [-0.025 to 0.023], Standard Error of Mean 0.012
Statistical Analysis 2: Comparison: Olmesartan (ARB) 40 mg PO Once Daily vs Placebo; Test type: Superiority or Other; p = 0.280, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Slope = 0.014, 95% CI 2-sided [-0.012 to 0.039], Standard Error of Mean 0.013
Statistical Analysis 3: Comparison: Alpha Lipoic Acid (ALA) 600 mg PO Twice Daily vs Placebo; Test type: Superiority or Other; p = 0.313, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Slope = 0.012, 95% CI 2-sided [-0.012 to 0.037], Standard Error of Mean 0.012

3. Other Pre Specified Outcome: AIM 2: Difference in FMD (Measure of Endothelial Function)
Description: Comparison of FMD (measure of endothelial function) between NGT, IGT and diabetes at baseline. FMD is a surrogate measure of endothelial function defined as the percent change in dilation of the brachial artery after cuff compression of arm compared to before cuff compression.
  No analysis was conducted due to under-recruitment.
Time Frame: Cross-sectional
Groups:
- Normal Glucose Tolerance (NGT): Normal fasting glucose (<100 mg/dl) and normal 2-hr glucose level (<140 mg/dl) after 75g OGTT
- Impaired Glucose Tolerance (IGT): After 75g OGTT:
  Fasting glucose <126 mg/dl and 2-hr glucose level 140-199 mg/dl
- Diabetes: After 75g OGTT:
  Fasting glucose >=126 mg/dl and 2-hr glucose level >=200 mg/dl
Arm/Group | Normal Glucose Tolerance (NGT) | Impaired Glucose Tolerance (IGT) | Diabetes
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Aspirin: Anti-inflammatory agent
- Olmesartan: Angiotensin receptor blocker (ARB)
- Alpha Lipoic Acid: Antioxidant
- Enrolled, But Not Yet Randomized: Enrolled into study, but not yet randomized to study medication
Arm/Group | Aspirin | Olmesartan | Alpha Lipoic Acid | Placebo | Enrolled, But Not Yet Randomized
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/17 | 1/14
Other Adverse Events (participants affected / at risk) | 0/18 | 1/18 | 0/17 | 0/17 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=18) | Olmesartan (N=18) | Alpha Lipoic Acid (N=17) | Placebo (N=17) | Enrolled, But Not Yet Randomized (N=14)
Cancer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pt was diagnosed with pancreatic cancer soon after enrollment, but before randomization to intervention group.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=18) | Olmesartan (N=18) | Alpha Lipoic Acid (N=17) | Placebo (N=17) | Enrolled, But Not Yet Randomized (N=14)
Reaction to nitroglycerin during FMD test (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — During baseline FMD testing, prior to actually starting study medication, a vasavagal response to NTG was developed.

LIMITATIONS AND CAVEATS:
Not fully powered due to under-enrollment and high drop-out rate. Higher than anticipated precision error of FMD measures. Possible Hawthorne effect with lifestyle changes. Short treatment period relative to long-term CVD risk in prediabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes